CLINICAL TRIAL: NCT06696612
Title: Dermoscopic Nail Changes in Vitiligo
Brief Title: Dermoscopy in Nails
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rehab Sotohy Ahmad Sotohy, Postgraduate student, Assiut University
Other Study IDs: Nail Dermoscopy
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Vitiligo; Healthy
MeSH Terms: conditions — Vitiligo | interventions — Dermoscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Dermoscopy — Dermoscopic examination of the nails

SUMMARY:
Study types and frequency of nail changes in patients with vitiligocompared to healthy subjects

DETAILED DESCRIPTION:
Dermoscopy is a noninvasive diagnostic tool that is currently being used for different skin lesions, several inflammatory & infectious diseases, and skin appendages disorders. ") In daily practice, dermoscopy may confirm clinical diagnosis and guides in the management of nail diseases, permitting a better visualization of symptoms. (2) Nail dermoscopy (Onychoscopy) was initially used only in the assessment of nail pigmentation, but now it is widely utilized for the evaluation of many nail disorders. (3) It enhances visible nail features; however, it can also help identify additional unique and fascinating features not visible to the naked eye. 2) Vitiligo is an acquired dyschromia of the skin in which there is loss of epidermal melanocytes The prevalence of vitiligo is approximately 0.1 - 2% worldwide. (5) Vitiligo is classified as segmental, acrofacial, generalized, and universal and less commonly mucosal and trichome.

Vitiligo has been described as a systemic disease. It has been associated with other autoimmune disorders as Diabetes (DM), Lupus, Psoriasis, Alopecia areata (AA), Hashimoto thyroiditis, and Gravesdisease.

Nails can show changes in association with many disorders such as renal, hepatic, pulmonary, autoimmune and collagen diseases. (67) Dermoscopic nail changes has been reported in several autoimmune disorders such as, in DM; longitudinal striations, pitting, onycholysis, & splinter hemorrhage, (® in AA; scaly cuticle, punctate leukonychia, oncholysis, &oncychoschizia®and in Collagen Vascular disorders; dilated capillaries, capillary dropout, and avascular areas. (10) To the best of our knowledge, dermoscopic nail changes in vitiligo haven't been reported yet. However, few studies had discussed clinical nail changes in vitiligo such as: (11) longitudinal ridging, absent lunula, leukonychia, pitting, in addition to less common nail changes such as flag sign and Terry's nails

ELIGIBILITY:
Inclusion Criteria:

* Age Adults patients 12-50 years old All types of vitiligo: Focal, generalized, acrofacial, segmental

Exclusion Criteria:

* patients older than 50 (because of aging's nail changes Patients with autoimmune disorders Patients using systemic medication for any reason including oral contraceptive pill

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Vitiligo patients attending dermatology outpatient clinic of Assiut University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Nail changes in Vitiligo | At enrollment
  Dermoscopic pictures of the nails